CLINICAL TRIAL: NCT02710916
Title: SD-OCT Multimodal Analysis in GLaucoma
Acronym: SOMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CHUBX 2015/20
Record Dates: First submitted 2016-03-04; First posted 2016-03-17 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Glaucoma; Ocular Hypertension; Eye Diseases
Keywords: Optical Coherence Tomography; Intraocular pressure; Optic Nerve Head; Nerve fiber layer; Bruch Membrane Opening -Minimum Rim Width
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- perimetric glaucoma patients (Sham Comparator)
  Interventions: Device: SD-OCT Spectralis
- preperimetric glaucoma patients (Active Comparator)
  Interventions: Device: SD-OCT Spectralis
- perimetric glaucoma control patients (Sham Comparator)
  Interventions: Device: SD-OCT Spectralis

INTERVENTIONS:
Device: SD-OCT Spectralis — All patients will undergo a complete ophthalmological examination with SD-OCT complete evaluation

SUMMARY:
Glaucoma is the first cause of irreversible blindness worldwide with more than 60 millions people affected in 2010. It is defined as a neurodegenerative disease characterized by a progressive loss of retinal ganglion cells (RGC), visual field deterioration and optic nerve excavation. Intraocular pressure (IOP) is the most common risk factor. Despite its severity, its impact on quality of life and an existing treatment that can delay visual field damages, there is no recommended strategy to screen the disease. Clinical evaluation of optic nerve head excavation performed either by ophthalmologists or glaucoma specialists is highly inter-observer dependent and limits its accuracy to diagnose glaucoma. Additionally, up to 30 to 40% of nerve fiber layer may be lost before detecting first visual field defects, thus making this tool not accurate enough for screening purposes.

Spectral-Domain Optical coherence tomography (SD-OCT) imaging technology allows precise and reproducible measurements of optic nerve head structures and retinal layers mainly related to the speed of acquisition and an axial resolution of 5 microns. New SD-OCT parameters have been developed to improve its diagnostic accuracy for glaucoma disease. The investigators therefore investigate performances of SD-OCT to discriminate glaucoma patients and controls. All subjects will undergo SD-OCT imaging (Spectralis™ OCT, Version 6.3, Heidelberg Engineering, Germany) and other study procedures in one single visit. All examinations performed on the subjects are non-significant risk.

ELIGIBILITY:
Inclusion Criteria: Normal Subjects

1. No history or evidence of retinal pathology or glaucoma
2. Normal Humphrey 24-2 Visual Field (VF) : A mean defect (MD), corrected pattern standard deviation (CPSD) within 95% limits of normal reference, and glaucoma hemifield test (GHT) within normal limits (97%).
3. Intraocular pressure < 21 mm Hg
4. Open angle (Shaffer's grading system)
5. Normal appearing Optic Nerve Hypoplasia (ONH) and Nerve Fiber Layer (NFL) : intact neuroretinal rim without peripapillary hemorrhages, notches, localized pallor, or NFL defect
6. Symmetric ONH between left and right eyes: Cup-to-Disc Ratio (CDR) difference < 0.2 in both vertical and horizontal dimensions

Inclusion Criteria: Perimetric Glaucoma

1. ONH or NFL defect visible on slit-lamp biomicroscopy defined as one of following:

   * diffuse or localized thinning of the rim
   * disc (splinter) hemorrhage
   * notch in the rim
   * vertical cup/disc ratio greater than the fellow eye by > 0.2
2. Consistent glaucomatous pattern on both qualifying Humphrey Swedish Interactive Threshold Algorithm (SITA) 24-2 VF meeting at least one of the following quantitative criteria for abnormality:

   * PSD outside normal limits (p < 0.05)
   * GHT outside normal limits (p < 0.01)

Inclusion Criteria: Pre-Perimetric Glaucoma (PPG)

PPG participants must have at least one eye meeting all of the following criteria:

1. ONH or NFL defect visible on slit-lamp biomicroscopy defined as one of following:

   * diffuse or localized thinning of the rim
   * disc (splinter) hemorrhage
   * notch in the rim
   * well-defined peripapillary NFL bundle defect.
   * inter-eye vertical CDR asymmetry > 0.2
2. Baseline VF not meeting the criteria for the PG group.
3. Risk factors for glaucoma, one of following:

   * Intraocular pressure > 21 mm Hg
   * Ethnics
   * Family history of glaucoma

Exclusion Criteria: All Groups

1. Age < 40
2. Refractive error of > +6.00 D or < -6.00 D (SE), +3,00 D for astigmatism
3. Diabetic retinopathy
4. Other diseases that may cause VF loss or optic disc abnormalities
5. Inability to clinically view or photograph the optic discs due to media opacity or poorly dilating pupil
6. Inability to perform reliably on automated VF testing
7. Insufficient quality of Spectralis OCT images (this is not determined until after Spectralis OCT examination, and is an unusual circumstance). Minimum requirements are:

   * Retina completely included in image frame,
   * Quality Score ≥ 15 in the stored mean images,
8. Refusal of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of Bruch's Membrane Opening Minimum Rim Width | 1 day
  Diagnostic accuracy of SD-OCT to discriminate perimetric, preperimetric glaucoma patients and control patients

SECONDARY OUTCOMES:
Evaluation of Retinal Nerve Fiber Layer Thickness | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University Bordeaux Hospital, Bordeaux, Aquitaine, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weinreb RN, Khaw PT. Primary open-angle glaucoma. Lancet. 2004 May 22;363(9422):1711-20. doi: 10.1016/S0140-6736(04)16257-0. PMID 15158634
- [Background] Klein BE, Klein R, Sponsel WE, Franke T, Cantor LB, Martone J, Menage MJ. Prevalence of glaucoma. The Beaver Dam Eye Study. Ophthalmology. 1992 Oct;99(10):1499-504. doi: 10.1016/s0161-6420(92)31774-9. PMID 1454314
- [Background] Sommer A, Tielsch JM, Katz J, Quigley HA, Gottsch JD, Javitt J, Singh K. Relationship between intraocular pressure and primary open angle glaucoma among white and black Americans. The Baltimore Eye Survey. Arch Ophthalmol. 1991 Aug;109(8):1090-5. doi: 10.1001/archopht.1991.01080080050026. PMID 1867550
- [Background] Leibowitz HM, Krueger DE, Maunder LR, Milton RC, Kini MM, Kahn HA, Nickerson RJ, Pool J, Colton TL, Ganley JP, Loewenstein JI, Dawber TR. The Framingham Eye Study monograph: An ophthalmological and epidemiological study of cataract, glaucoma, diabetic retinopathy, macular degeneration, and visual acuity in a general population of 2631 adults, 1973-1975. Surv Ophthalmol. 1980 May-Jun;24(Suppl):335-610. PMID 7444756
- [Background] Leung CK, Lam S, Weinreb RN, Liu S, Ye C, Liu L, He J, Lai GW, Li T, Lam DS. Retinal nerve fiber layer imaging with spectral-domain optical coherence tomography: analysis of the retinal nerve fiber layer map for glaucoma detection. Ophthalmology. 2010 Sep;117(9):1684-91. doi: 10.1016/j.ophtha.2010.01.026. Epub 2010 Jul 21. PMID 20663563
- [Background] Leung CK, Choi N, Weinreb RN, Liu S, Ye C, Liu L, Lai GW, Lau J, Lam DS. Retinal nerve fiber layer imaging with spectral-domain optical coherence tomography: pattern of RNFL defects in glaucoma. Ophthalmology. 2010 Dec;117(12):2337-44. doi: 10.1016/j.ophtha.2010.04.002. Epub 2010 Aug 3. PMID 20678802
- [Background] Windisch BK, Harasymowycz PJ, See JL, Chauhan BC, Belliveau AC, Hutchison DM, Nicolela MT. Comparison between confocal scanning laser tomography, scanning laser polarimetry and optical coherence tomography on the ability to detect localised retinal nerve fibre layer defects in glaucoma patients. Br J Ophthalmol. 2009 Feb;93(2):225-30. doi: 10.1136/bjo.2008.141945. Epub 2008 Sep 2. PMID 18765430
- [Background] Alasil T, Wang K, Yu F, Field MG, Lee H, Baniasadi N, de Boer JF, Coleman AL, Chen TC. Correlation of retinal nerve fiber layer thickness and visual fields in glaucoma: a broken stick model. Am J Ophthalmol. 2014 May;157(5):953-59. doi: 10.1016/j.ajo.2014.01.014. Epub 2014 Jan 30. PMID 24487047
- [Background] Horn FK, Mardin CY, Laemmer R, Baleanu D, Juenemann AM, Kruse FE, Tornow RP. Correlation between local glaucomatous visual field defects and loss of nerve fiber layer thickness measured with polarimetry and spectral domain OCT. Invest Ophthalmol Vis Sci. 2009 May;50(5):1971-7. doi: 10.1167/iovs.08-2405. Epub 2009 Jan 17. PMID 19151389
- [Background] Leaney J, Healey PR, Lee M, Graham SL. Correlation of structural retinal nerve fibre layer parameters and functional measures using Heidelberg Retinal Tomography and Spectralis spectral domain optical coherence tomography at different levels of glaucoma severity. Clin Exp Ophthalmol. 2012 Nov;40(8):802-12. doi: 10.1111/j.1442-9071.2012.02807.x. Epub 2012 Jul 2. PMID 22594488
- [Background] Chauhan BC, O'Leary N, AlMobarak FA, Reis ASC, Yang H, Sharpe GP, Hutchison DM, Nicolela MT, Burgoyne CF. Enhanced detection of open-angle glaucoma with an anatomically accurate optical coherence tomography-derived neuroretinal rim parameter. Ophthalmology. 2013 Mar;120(3):535-543. doi: 10.1016/j.ophtha.2012.09.055. Epub 2012 Dec 23. PMID 23265804
- [Background] Bussel II, Wollstein G, Schuman JS. OCT for glaucoma diagnosis, screening and detection of glaucoma progression. Br J Ophthalmol. 2014 Jul;98 Suppl 2(Suppl 2):ii15-9. doi: 10.1136/bjophthalmol-2013-304326. Epub 2013 Dec 19. PMID 24357497
- [Background] Almobarak FA, O'Leary N, Reis AS, Sharpe GP, Hutchison DM, Nicolela MT, Chauhan BC. Automated segmentation of optic nerve head structures with optical coherence tomography. Invest Ophthalmol Vis Sci. 2014 Feb 26;55(2):1161-8. doi: 10.1167/iovs.13-13310. PMID 24474272
- [Background] Wu H, de Boer JF, Chen TC. Diagnostic capability of spectral-domain optical coherence tomography for glaucoma. Am J Ophthalmol. 2012 May;153(5):815-826.e2. doi: 10.1016/j.ajo.2011.09.032. Epub 2012 Jan 20. PMID 22265147
- [Background] Wu H, de Boer JF, Chen TC. Reproducibility of retinal nerve fiber layer thickness measurements using spectral domain optical coherence tomography. J Glaucoma. 2011 Oct;20(8):470-6. doi: 10.1097/IJG.0b013e3181f3eb64. PMID 20852437
- [Background] Alasil T, Wang K, Keane PA, Lee H, Baniasadi N, de Boer JF, Chen TC. Analysis of normal retinal nerve fiber layer thickness by age, sex, and race using spectral domain optical coherence tomography. J Glaucoma. 2013 Sep;22(7):532-41. doi: 10.1097/IJG.0b013e318255bb4a. PMID 22549477
- [Background] Wessel JM, Horn FK, Tornow RP, Schmid M, Mardin CY, Kruse FE, Juenemann AG, Laemmer R. Longitudinal analysis of progression in glaucoma using spectral-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2013 May 1;54(5):3613-20. doi: 10.1167/iovs.12-9786. PMID 23633657
- [Background] Langenegger SJ, Funk J, Toteberg-Harms M. Reproducibility of retinal nerve fiber layer thickness measurements using the eye tracker and the retest function of Spectralis SD-OCT in glaucomatous and healthy control eyes. Invest Ophthalmol Vis Sci. 2011 May 18;52(6):3338-44. doi: 10.1167/iovs.10-6611. PMID 21330656
- [Background] El Chehab H, Delbarre M, Marechal M, Rosenberg R, Marill AF, Fenolland JR, Renard JP. [New neuroretinal rim analysis with spectral domain optical coherence tomography, Spectralis (Heidelberg Engineering, Germany). Preliminary study]. J Fr Ophtalmol. 2015 Jan;38(1):46-52. doi: 10.1016/j.jfo.2014.10.004. Epub 2015 Jan 6. French. PMID 25575418
- [Background] Strouthidis NG, Yang H, Fortune B, Downs JC, Burgoyne CF. Detection of optic nerve head neural canal opening within histomorphometric and spectral domain optical coherence tomography data sets. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):214-23. doi: 10.1167/iovs.08-2302. Epub 2008 Aug 8. PMID 18689697
- [Background] Strouthidis NG, Grimm J, Williams GA, Cull GA, Wilson DJ, Burgoyne CF. A comparison of optic nerve head morphology viewed by spectral domain optical coherence tomography and by serial histology. Invest Ophthalmol Vis Sci. 2010 Mar;51(3):1464-74. doi: 10.1167/iovs.09-3984. Epub 2009 Oct 29. PMID 19875649
- [Background] Strouthidis NG, Yang H, Downs JC, Burgoyne CF. Comparison of clinical and three-dimensional histomorphometric optic disc margin anatomy. Invest Ophthalmol Vis Sci. 2009 May;50(5):2165-74. doi: 10.1167/iovs.08-2786. Epub 2009 Jan 10. PMID 19136694
- [Background] Downs JC, Roberts MD, Burgoyne CF. Mechanical environment of the optic nerve head in glaucoma. Optom Vis Sci. 2008 Jun;85(6):425-35. doi: 10.1097/OPX.0b013e31817841cb. PMID 18521012
- [Background] Burgoyne CF, Downs JC, Bellezza AJ, Suh JK, Hart RT. The optic nerve head as a biomechanical structure: a new paradigm for understanding the role of IOP-related stress and strain in the pathophysiology of glaucomatous optic nerve head damage. Prog Retin Eye Res. 2005 Jan;24(1):39-73. doi: 10.1016/j.preteyeres.2004.06.001. PMID 15555526
- [Background] Burgoyne CF, Morrison JC. The anatomy and pathophysiology of the optic nerve head in glaucoma. J Glaucoma. 2001 Oct;10(5 Suppl 1):S16-8. doi: 10.1097/00061198-200110001-00007. No abstract available. PMID 11890263
- [Background] Johnstone J, Fazio M, Rojananuangnit K, Smith B, Clark M, Downs C, Owsley C, Girard MJ, Mari JM, Girkin CA. Variation of the axial location of Bruch's membrane opening with age, choroidal thickness, and race. Invest Ophthalmol Vis Sci. 2014 Mar 28;55(3):2004-9. doi: 10.1167/iovs.13-12937. PMID 24595390